CLINICAL TRIAL: NCT00488085
Title: Crohn's Disease, Obesity and Disease Severity
Acronym: CROHN_OBESE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Other Study IDs: TASMC-07-ID-173-CTIL
Record Dates: First submitted 2007-06-17; First posted 2007-06-19 (Estimated); Last update posted 2007-06-19 (Estimated); Status verified 2007-03

CONDITIONS: Crohn's Disease, Obesity
Keywords: Crohn's disease, obesity, REE, body composition, fat absorption
MeSH Terms: conditions — Crohn Disease; Obesity

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of our study is to suggest possible underlying mechanisms for the observed clinical differences in disease severity and behavior of overweight and obese patients with crohn's disease(BMI > 25 kg/m²)as compare to non-obese crohn's patients with a normal or low weight ( BMI ≤ 25) by measuring metabolic\nutritional variables and cytokine levels.

DETAILED DESCRIPTION:
Crohn's disease (CD) is a chronic intestinal disorder of unknown etiology that may involve any part of the gastrointestinal tract. The small bowel is involved in 70% of CD patients.

Undernutrition expressed in low body mass index (BMI) <18.5 kg/m², is a common presentation and has been reported in 65-75% of these patients. Possible pathogenic mechanisms include inadequate dietary intake ,increased energy expenditure, nutrient malabsorption and intestinal losses. We have studied recently these three important components of energy balance of underweight crohn's patients and found that nutrient malabsorption may play a role.

Although the majority of crohn's disease patients are undernourished , some of them are surprisingly obese and their symptoms seem be more severe; Blain A et al. have reported recently that obesity in CD has been associated with more frequent anoperineal complications and a more marked disease activity. Hass J et al have found that overweight CD patients require earlier surgical intervention and perhaps more aggressive medical therapy. Notwithstanding, the characteristics of CD and possible underlying pathophysiological mechanisms in obese patients have not been studied yet.

Mesenteric hypertrophied fat commonly called "creeping fat is a common feature of crohn's disease and has been reported to correlate with ulceration, stricture formation and transmural inflammation. It is a matter of debate whether the development of creeping fat is a causative or secondary phenomenon ,but there is increasing body of evidence that suggest that mesenteric adipose tissue plays an active role in the pathogenesis of creeping fat and mesenteric inflammation by pro-inflammatory and anti-inflammatory adipocytokines.

Recently there is more recognition that adipose tissue is not a passive connective tissue merely storing fat but an activeendocrine organ which participates in numerous physiological and pathophysiological processes with variety of secretory products designated adipocytokines that regulate metabolic processes in an endocrine ,paracrine and autocrine manner Moreover, Obesity is increasingly being recognized as a risk factor for a number of gastrointestinal conditions as well as being characterized by a chronic, systemic low-grade state of inflammation per se. Biomarkers of inflammation, such as the leukocyte count, tumor necrosis factor-alpha (TNF-alpha), interleukin 6 (IL-6), and C-reactive protein, are increased in obesity and have been related to insulin resistance and the metabolic syndrome.

ELIGIBILITY:
Inclusion criteria:

1. Age > 18 years
2. No other chronic diseases except obesity -related (NAFLD, NASH etc).
3. Stable (LESS THAN 10% CHANGE) body weight during the 3 months preceding the study.

Exclusion criteria:

1. Patients with internal fistulae (perianal disease allowed)
2. Ileostomy or colostomy
3. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-06; Study Completion 2007-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Nachum Vaisman, Prof., Study Director — The Unit of Clinical Nutrition
Locations (1):
- The Unit of Clinical Nutrition, Tel Aviv, Israel